CLINICAL TRIAL: NCT04356950
Title: Analysis of the Coagulopathy Developed by COVID-19 Infected Patients: Thrombin Generation Potential in COVID-19 Infected Patients
Brief Title: Analysis of the Coagulopathy Developed by COVID-19 Infected Patients
Acronym: COVID-TGT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2020/JCG-01; 2020-A01068-31 (Other: ANSM)
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-09

CONDITIONS: Sepsis; Blood Coagulation Disorders; Thrombin; Disseminated Intravascular Coagulation; COVID-19
Keywords: coagulation; survival; thrombin generation test
MeSH Terms: conditions — Sepsis; Blood Coagulation Disorders; Disseminated Intravascular Coagulation; COVID-19; Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thrombin generation test assay — lag time, initial velocity, time-to-peak, thrombin peak, total thrombin generation time, extrinsic thrombin potential (ETP). Crude quantitative values and relative values (%, by reference to the one obtained with an invariant reference plasma). Both without the addition of purified thrombomodulin (TM-) and with the addition of purified thrombomodulin (TM+). The ability of TM to inhibit thrombin generation will be calculated as follows: [ETP (%)(TM+) / ETP (%)(TM-)].
Other: Fibrin generation markers assays — D-dimers (coagulation plus fibrinolysis), soluble fibrin monomers (coagulation only)

SUMMARY:
Increased D-dimers at admission of COVID-19 infected patients entering hospital due to a severe disease is a risk factor for death. Understanding this acquired coagulopathy is a prerequisite before specific interventional studies. The study investigators aim to apply a normalized and automated thrombin generation test (TGT), developed for testing the thrombotic risk (triggered by 5 pM Tissue Factor, with a purified thrombomodulin (TM) challenge) and to study its association with survival.

DETAILED DESCRIPTION:
Accumulating data describe, in COVID-19 severely infected patients necessitating hospitalized medical support, the development of an acquired coagulopathy, from a sepsis-induced coagulopathy to an overt-DIC, which is a strong risk factor for death. Understanding this coagulopathy is a prerequisite before specific interventional studies. Conventional coagulation tests, like prothrombin time PT and aPTT, only reflect 5% of the total thrombin generation and are insensitive to the patients' natural anticoagulants. The investigators thus wish to analyze the coagulopathy of SARS-CoV-2 using a global analytical test reflecting the full complexity of thrombin generation then inhibition, the thrombin generation test (TGT), in its version designed to analyze the thrombotic risk (initiation by an intermediate concentration of human Tissue: 5 pM), in its fully automated and standardized technical version. This test analyzes not only the generation of thrombin and its various informative phases (initiation phase, propagation phase culminating at the peak of formation, inhibition phase with natural anticoagulants) but also the capacity for an exogenous addition of purified thrombomodulin (TM), which quantifies the anticoagulant activity of the patient's protein C activated by thrombin, to inhibit this generation of thrombin.

The aim is to assay this TGT version in a centralized way, on the patients' plasma obtained at hospital admission, just after checking the positive COVID-19 testing , together with the traditional blood tests including platelet counts, PT, D-dimers (DDi) and soluble fibrin monomers (FMs). The various quantitative biological parameters describing the results of the TGT assay, together with relevant covariates, will be tested using multivariate analysis for their capacity to be risk factors for clinically-relevant qualitative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with SARS-CoV-2 infection entering hospitalization with or without resuscitation
* The patient (or their carer) must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Pregnant or breastfeeding patient
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Thrombotic events during treatment: flare-up of venous thromboembolism, flare-up of atherothrombosis.
* Long-term anticoagulant treatment (anti-vitamin K, direct oral anticoagulant).
* Chronic anti-aggregation treatment.
* Pre-existing constitutive or acquired known coagulation pathology: hemorrhagic diseases (thrombocytopenia, thrombocytopathy, hemophilia, von Willebrand's disease, hemorrhagiparous factor deficiency), and for thrombophilia (deficits in antithrombin, protein C or S , Factor V Leiden or Prothrombin 20201A mutation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients hospitalized for SARS-CoV-2 infection with symptomatology / severity requiring hospital treatment.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
28-day survival rate | 1 month
  Death yes/no during hopstilization, 28 days after admittence
Absolute thrombin generation test latent period | Day 0
  Seconds; without (TM-) and with (TM+) purified thrombomodulin
Relative thrombin generation test latent period compared to reference plasma | Day 0
  %; without (TM-) and with (TM+) purified thrombomodulin
Absolute thrombin generation test initial velocity | Day 0
  nmol/s; without (TM-) and with (TM+) purified thrombomodulin
Relative thrombin generation test initial velocity compared to reference plasma | Day 0
  %; without (TM-) and with (TM+) purified thrombomodulin
Relative thrombin generation test peak thrombin compared to reference plasma | Day 0
  %; without (TM-) and with (TM+) purified thrombomodulin
Absolute thrombin generation test peak thrombin | Day 0
  nmol/L; without (TM-) and with (TM+) purified thrombomodulin
Absolute thrombin generation test peak thrombin time | Day 0
  Seconds; without (TM-) and with (TM+) purified thrombomodulin
Relative thrombin generation test peak thrombin time compared to reference plasma | Day 0
  %; without (TM-) and with (TM+) purified thrombomodulin
Absolute thrombin generation test total thrombin generation time | Day 0
  seconds; without (TM-) and with (TM+) purified thrombomodulin
Relative thrombin generation test total thrombin generation time compared to reference plasma | Day 0
  %; without (TM-) and with (TM+) purified thrombomodulin
Absolute thrombin generation test endogenous thrombin potential | Day 0
  Seconds; without (TM-) and with (TM+) purified thrombomodulin
Relative thrombin generation test endogenous thrombin potential compared to reference plasma | Day 0
  %; without (TM-) and with (TM+) purified thrombomodulin

SECONDARY OUTCOMES:
3-month survival rate | 3 months
  Death yes/no
Transfer to intensive care unit during hospitalization | 3 months
  Yes/no
Thrombotic complication during hospitalization | 3 months
  Yes/no (deep vein thrombosis, pulmonary embolism, atherothrombosis flare, arterial thrombosis)
Plasma concentrations of D-dimers | Day 0
  µg / L, assayed by automated enzyme linked fluorescent assay (Vidas® D-dimers Exclusion ™ II)
Plasma concentrations of soluble fibrin monomers | Day 0
  mg / L, measured by automated immunoagglutination (STA®-Liatest® FM)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Gris, Principal Investigator — CHU Nimes
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CHU de Limoges, Limoges
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes

REFERENCES:
- [Result] Gris JC, Guillotin F, Dos Santos TP, Chea M, Loubet P, Laureillard D, Sotto A, Muller L, Barbar SD, Roger C, Lefrant JY, Jung B, Klouche K, Mura T, Quere I, Perez-Martin A. Prognostic value of an automated thrombin generation assay in COVID-19 patients entering hospital: A multicentric, prospective observational study. Thromb Res. 2023 Feb;222:85-95. doi: 10.1016/j.thromres.2022.12.019. Epub 2023 Jan 2. PMID 36608393